CLINICAL TRIAL: NCT06010667
Title: A Prospective, Randomized Controlled Study of Cyclophosphamide, Bevacizumab With or Without Envafolimab in Recurrent Epithelial Ovarian Cancer (EOC), Fallopian Tube Cancer, and Primary Peritoneal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhengmao ZHANG
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — envafolimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EBC: cyclophosphamide and bevacizumab in combination with Envafolimab
  Interventions: Drug: Envafolimab
- BC: cyclophosphamide in combination with Envafolimab

INTERVENTIONS:
Drug: Envafolimab — With or without Envafolimab
  Groups: EBC

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of cyclophosphamide and bevacizumab in combination with Envafolimab in the treatment of recurrent epithelial ovarian cancer (EOC), fallopian tube cancer, and primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years Histologically or pathologically confirmed epithelial ovarian cancer (EOC), fallopian tube cancer, primary peritoneal cancer Patients with recurrent ovarian, fallopian tube, and primary peritoneal cancer following platinum-based chemotherapy measurable lesions (according to RECIST 1.1 criteria, non-lymph node lesions CT scan long diameter ≥ 10 mm, lymph node lesions CT scan short diameter ≥ 15 mm) ECOG PS score: 0 - 1;

Exclusion Criteria:

* Subject has prior or concurrent other malignancy Prior treatment with other PD-L1/PD-L1 inhibitors cannot be enrolled; Subject has known previous hypersensitivity to macromolecular protein preparations or applied drug components

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: epithelial ovarian cancer (EOC), fallopian tube cancer, primary peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate;ORR | 2years
  CR+PR

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No